CLINICAL TRIAL: NCT04026698
Title: Implementing an Intervention to Foster Meaningful Engagement and Shared Decision-making in Long-term Care: A Mixed Methods Approach
Brief Title: Implementing an Intervention to Foster Resident and Family Engagement in Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Lisa Cranley, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 36220
Record Dates: First submitted 2019-07-04; First posted 2019-07-19 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Quality of Life

STUDY DESIGN:
Intervention Model Description: This intervention study has a single group of participants who will receive the intervention. There is no control group or randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resident and Family Engagement Intervention. (Experimental): The intervention has three components: leadership coaching for managers, administrators/ directors of care in long-term care settings; a one-day in-person training session for staff and managers; and resident and family led huddles (brief, 15 minute meetings) with staff.
  Interventions: Behavioral: Resident and Family Engagement Intervention

INTERVENTIONS:
Behavioral: Resident and Family Engagement Intervention — The leadership coaching component targets managers, administrators/ directors of care in long-term care settings. These sessions involve selecting a subset of relevant performance outcomes from the quality improvement plan that align with leadership vision and priorities for staff performance which leaders can monitor, reinforce and encourage.
  The education component involves a one-day in-person training session for staff and managers on communication strategies and ways to engage family and residents in care planning, and includes follow-up visits.
  The huddle component involves a series of resident and family led huddles (brief, 15 minute meetings) to discuss a care related topic with staff to foster proactive communication and information sharing. Resident-family dyads will participate in the huddles, along with the staff and management team who received the training. The huddles will be scheduled for 15 minutes once/month for up to 3 months.

SUMMARY:
This study is a pilot test of an intervention to engage residents and their family and the healthcare team in a collaborative approach to decisions about care planning in long-term care. The intervention includes leadership coaching with the management team, an educational bundle that includes a one-day education session for staff and managers on communication strategies and ways to engage family and residents in care planning and follow-up visits, and a series of resident and family led huddles (brief, 15 minute meetings) to discuss a care related topic with staff to foster proactive communication and information sharing for care planning.

DETAILED DESCRIPTION:
This study is a pilot test of an intervention to engage residents and their family and the healthcare team in a collaborative approach to decisions about care planning in long-term care. The intervention includes leadership coaching with the management team, an educational bundle that includes a one-day education session for staff and managers on communication strategies and ways to engage family and residents in care planning and follow-up visits, and a series of resident and family led huddles (brief, 15 minute meetings) to discuss a care related topic with staff to foster proactive communication and information sharing and care planning.

The study aims are to describe the feasibility and acceptability of the resident and family engagement intervention, and to evaluate the following outcomes: resident quality of life, resident and family satisfaction with care, and staff quality of work life. The investigators aim to recruit 20 staff, the leadership team, and 12 resident-family dyads from four long-term care facilities who will receive the intervention and complete the survey measures. The expected outcome from this study is an increased understanding of how to engage residents and family in care decisions impacting quality of life.

Amendment: Due to the COVID-19 pandemic, the anticipated sample size is smaller and as a result, our outcomes will be explored qualitatively through interviews.

ELIGIBILITY:
Inclusion Criteria for Residents:

* residents who can communicate in English
* residents (aged 65 or older) who have a visiting family member who is their substitute decision maker- both the resident and their family member will participate in the huddles

Exclusion Criteria:

* residents with severe cognitive impairment
* residents who do not speak English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Quality of life- a change is being assessed | Pre-intervention and post-intervention- within 3 months after intervention completion
  The dementia quality of life DEMQOL (28-items) and DEMQOL-Proxy (31-items) are measures that assess health-related quality of life of people with dementia. The questions are interviewer-administered to obtain self (person with dementia) and caregiver perspectives. Response options range from 1=a lot to 4=not at all (with higher scores indicating a higher perceived health-related quality of life). A total score is calculated by summing scores from the 28 items (minimum score 28, maximum score 112).

SECONDARY OUTCOMES:
Resident satisfaction with care- a change is being assessed | Pre-intervention and post-intervention- within 3 months after intervention completion
  Resident satisfaction with care will be assessed using the Resident Satisfaction with the Nursing Home questionnaire, a 29-item measure that has been used with residents with cognitive impairment. The questions are interviewer-administered to obtain self-reported data from the resident using Yes/No response options (with a Yes response indicating satisfaction).
Family satisfaction with resident care- a change is being assessed | Pre-intervention and post-intervention- within 3 months after intervention completion
  Family satisfaction with resident care will be assessed using the Nursing Facility Family Satisfaction Questionnaire, a 20-item measure that uses a visual analogue scale ranging from 1 (very poor) to 10 (excellent).
Staff quality of work life- a change is being assessed | Pre-intervention and post-intervention- within 3 months after intervention completion
  Staff quality of work life will be assessed using a 16-item need-satisfaction measure on a five-point Likert scale ranging from 1=strongly disagree to 5=strongly agree (with higher scores indicating a higher perception of quality of work life).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Cranley, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cranley LA, McGillis Hall L, Duggleby W, Helfenbaum S, Galessiere D, Meyer RM, Sivakumaran G, Just D, MacEachern L, McGilton KS. Resident- and family-led huddles for collaborative care planning in long-term care: a feasibility study. Innov Aging. 2025 Oct 23;9(11):igaf116. doi: 10.1093/geroni/igaf116. eCollection 2025. PMID 41334049